CLINICAL TRIAL: NCT02761343
Title: MRI Assessment of Arrythmia Ablation Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Charles Berul, MD, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4065; contract (Other: NIH)
Record Dates: First submitted 2016-04-25; First posted 2016-05-04 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Ventricular Tachycardia; Cardiac Arrhythmia
Keywords: cardiac arrhythmia; cardiac ablation; congenital cardiac disease; cardiac ablation lesions under Magnetic Resonance imaging
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI scan (Other): Post ablation MRI scan will be performed for all subjects who are clinically stable.
  Interventions: Other: MRI scan

INTERVENTIONS:
Other: MRI scan — Following the clinically indicated cardiac ablation procedure, a post ablation MRI scan will be performed.

SUMMARY:
This study will evaluate the feasibility of visualization and characterization of arrhythmia ablation lesions by MRI immediately following standard ablation techniques. The appearance of the ablation lesion will be correlated with clinical outcomes and risk of arrhythmia recurrence.

DETAILED DESCRIPTION:
Children's National Heart Institute (CNHI) with major contractual support from the National Institutes of Health / National Heart, Lung and Blood Institute has installed a combined X-ray / Magnetic Resonance Imaging cardiac catheterization lab suite allowing for experts in the fields of cardiac MRI, interventional cardiac MRI and clinical pediatric interventional electrophysiology to work together to make substantial advancements in the development of novel techniques and applications to reach the goal of improved survival and care for the congenital heart disease population. The CNHI X-ray/MRI suite will allow for streamlined transfer of patients from fluoroscopy directly to the MRI scanner under the same sedation thereby allowing for immediate post procedure imaging and minimizing risk to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from any patient willing to participate who is undergoing an electrophysiology study with potential for arrhythmia ablation
* Written informed assent, if applicable

Exclusion Criteria:

* Women who are pregnant
* Women who are nursing and who do not plan to discard breast milk for 24 hours
* Patients with a contraindication to MRI scanning will be excluded. These contraindications include patients with the following devices:

  * Central nervous system aneurysm clips
  * Implanted neural stimulator
  * Implanted cardiac pacemaker or defibrillator which are not MR safe or MR conditional according to the manufacturer
  * Cochlear implant
  * Ocular foreign body (e.g. metal shavings)
  * Implanted Insulin pump
  * Metal shrapnel or bullet.
  * Any intracardiac or intravascular device that is not MR safe or MR conditional according to the manufacturer based on both material and timing of device placement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
The number of participants following ablation procedure who: a). have an arrythmia reoccurrence, b). require a repeat ablation procedure, and c). require treatment for arrhythmia management | Post ablation up to 5 years

SECONDARY OUTCOMES:
To measure the size of the ablation lesion on cardiac MR imaging | At the end of each ablation procedure through study completion, up to 5 years.
The number of post ablation MR images with a visible lesion. | At the end of each ablation procedure through study completion, up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Berul, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mondesert B, Abadir S, Khairy P. Arrhythmias in adult congenital heart disease: the year in review. Curr Opin Cardiol. 2013 May;28(3):354-9. doi: 10.1097/HCO.0b013e32835fb7c2. PMID 23511123
- [Background] Yap SC, Harris L, Silversides CK, Downar E, Chauhan VS. Outcome of intra-atrial re-entrant tachycardia catheter ablation in adults with congenital heart disease: negative impact of age and complex atrial surgery. J Am Coll Cardiol. 2010 Nov 2;56(19):1589-96. doi: 10.1016/j.jacc.2010.04.061. PMID 21029876
- [Background] Melby SJ, Lee AM, Zierer A, Kaiser SP, Livhits MJ, Boineau JP, Schuessler RB, Damiano RJ Jr. Atrial fibrillation propagates through gaps in ablation lines: implications for ablative treatment of atrial fibrillation. Heart Rhythm. 2008 Sep;5(9):1296-301. doi: 10.1016/j.hrthm.2008.06.009. Epub 2008 Jun 10. PMID 18774106
- [Background] Reddy VY, Schmidt EJ, Holmvang G, Fung M. Arrhythmia recurrence after atrial fibrillation ablation: can magnetic resonance imaging identify gaps in atrial ablation lines? J Cardiovasc Electrophysiol. 2008 Apr;19(4):434-7. doi: 10.1111/j.1540-8167.2007.01055.x. Epub 2007 Dec 20. PMID 18179530
- [Background] Ratnayaka K, Faranesh AZ, Hansen MS, Stine AM, Halabi M, Barbash IM, Schenke WH, Wright VJ, Grant LP, Kellman P, Kocaturk O, Lederman RJ. Real-time MRI-guided right heart catheterization in adults using passive catheters. Eur Heart J. 2013 Feb;34(5):380-9. doi: 10.1093/eurheartj/ehs189. Epub 2012 Aug 1. PMID 22855740
- [Background] Razavi R, Hill DL, Keevil SF, Miquel ME, Muthurangu V, Hegde S, Rhode K, Barnett M, van Vaals J, Hawkes DJ, Baker E. Cardiac catheterisation guided by MRI in children and adults with congenital heart disease. Lancet. 2003 Dec 6;362(9399):1877-82. doi: 10.1016/S0140-6736(03)14956-2. PMID 14667742
- [Background] Nazarian S, Kolandaivelu A, Zviman MM, Meininger GR, Kato R, Susil RC, Roguin A, Dickfeld TL, Ashikaga H, Calkins H, Berger RD, Bluemke DA, Lardo AC, Halperin HR. Feasibility of real-time magnetic resonance imaging for catheter guidance in electrophysiology studies. Circulation. 2008 Jul 15;118(3):223-9. doi: 10.1161/CIRCULATIONAHA.107.742452. Epub 2008 Jun 23. PMID 18574048
- [Background] Faddis MN, Chen J, Osborn J, Talcott M, Cain ME, Lindsay BD. Magnetic guidance system for cardiac electrophysiology: a prospective trial of safety and efficacy in humans. J Am Coll Cardiol. 2003 Dec 3;42(11):1952-8. doi: 10.1016/j.jacc.2003.07.023. PMID 14662258
- [Background] Ector J, De Buck S, Adams J, Dymarkowski S, Bogaert J, Maes F, Heidbuchel H. Cardiac three-dimensional magnetic resonance imaging and fluoroscopy merging: a new approach for electroanatomic mapping to assist catheter ablation. Circulation. 2005 Dec 13;112(24):3769-76. doi: 10.1161/CIRCULATIONAHA.105.565002. Epub 2005 Dec 5. PMID 16330683
- [Background] Kettering K, Greil GF, Fenchel M, Kramer U, Weig HJ, Busch M, Miller S, Sieverding L, Laszlo R, Schreieck J. Catheter ablation of atrial fibrillation using the Navx-/Ensite-system and a CT-/MRI-guided approach. Clin Res Cardiol. 2009 May;98(5):285-96. doi: 10.1007/s00392-009-0001-9. Epub 2009 Mar 13. PMID 19283334
- [Background] Sasaki T, Miller CF, Hansford R, Yang J, Caffo BS, Zviman MM, Henrikson CA, Marine JE, Spragg D, Cheng A, Tandri H, Sinha S, Kolandaivelu A, Zimmerman SL, Bluemke DA, Tomaselli GF, Berger RD, Calkins H, Halperin HR, Nazarian S. Myocardial structural associations with local electrograms: a study of postinfarct ventricular tachycardia pathophysiology and magnetic resonance-based noninvasive mapping. Circ Arrhythm Electrophysiol. 2012 Dec;5(6):1081-90. doi: 10.1161/CIRCEP.112.970699. Epub 2012 Nov 13. PMID 23149263
- [Background] Godeschalk-Slagboom CJ, van der Geest RJ, Zeppenfeld K, Botha CP. Cardiac MRI visualization for ventricular tachycardia ablation. Int J Comput Assist Radiol Surg. 2012 Sep;7(5):753-67. doi: 10.1007/s11548-012-0776-4. Epub 2012 Jul 3. PMID 22752391
- [Background] Dickfeld T, Tian J, Ahmad G, Jimenez A, Turgeman A, Kuk R, Peters M, Saliaris A, Saba M, Shorofsky S, Jeudy J. MRI-Guided ventricular tachycardia ablation: integration of late gadolinium-enhanced 3D scar in patients with implantable cardioverter-defibrillators. Circ Arrhythm Electrophysiol. 2011 Apr;4(2):172-84. doi: 10.1161/CIRCEP.110.958744. Epub 2011 Jan 26. PMID 21270103
- [Background] Yokokawa M, Mueller G, Bogun F. Role of imaging in ablation therapy of ventricular arrhythmias. Focus on cardiac magnetic resonance imaging. Circ J. 2012;76(6):1292-8. doi: 10.1253/circj.cj-12-0544. Epub 2012 May 22. PMID 22739077
- [Background] Nazarian S, Bluemke DA, Halperin HR. Applications of cardiac magnetic resonance in electrophysiology. Circ Arrhythm Electrophysiol. 2009 Feb;2(1):63-71. doi: 10.1161/CIRCEP.108.811562. PMID 19808444
- [Background] Mahnkopf C, Halbfass P, Turschner O, Brachmann J. [Use of cardiac MRI in the field of electrophysiology. Present status and future aspects]. Herzschrittmacherther Elektrophysiol. 2012 Dec;23(4):275-80. doi: 10.1007/s00399-012-0238-2. Epub 2012 Nov 7. German. PMID 23132745
- [Background] Kleinerman RA. Cancer risks following diagnostic and therapeutic radiation exposure in children. Pediatr Radiol. 2006 Sep;36 Suppl 2(Suppl 2):121-5. doi: 10.1007/s00247-006-0191-5. PMID 16862418
- [Background] Andreassi MG, Ait-Ali L, Botto N, Manfredi S, Mottola G, Picano E. Cardiac catheterization and long-term chromosomal damage in children with congenital heart disease. Eur Heart J. 2006 Nov;27(22):2703-8. doi: 10.1093/eurheartj/ehl014. Epub 2006 May 22. PMID 16717079
- [Background] Beels L, Bacher K, De Wolf D, Werbrouck J, Thierens H. gamma-H2AX foci as a biomarker for patient X-ray exposure in pediatric cardiac catheterization: are we underestimating radiation risks? Circulation. 2009 Nov 10;120(19):1903-9. doi: 10.1161/CIRCULATIONAHA.109.880385. Epub 2009 Oct 26. PMID 19858412
- [Background] Lima JA, Desai MY. Cardiovascular magnetic resonance imaging: current and emerging applications. J Am Coll Cardiol. 2004 Sep 15;44(6):1164-71. doi: 10.1016/j.jacc.2004.06.033. PMID 15364314
- [Background] Gupta S, Desjardins B, Baman T, Ilg K, Good E, Crawford T, Oral H, Pelosi F, Chugh A, Morady F, Bogun F. Delayed-enhanced MR scar imaging and intraprocedural registration into an electroanatomical mapping system in post-infarction patients. JACC Cardiovasc Imaging. 2012 Feb;5(2):207-10. doi: 10.1016/j.jcmg.2011.08.021. PMID 22340829
- [Background] Obeyesekere MN. MR scar imaging and intraprocedural registration into an electroanatomic mapping system in post-MI patients. JACC Cardiovasc Imaging. 2012 Aug;5(8):854; author reply 854-5. doi: 10.1016/j.jcmg.2012.05.010. No abstract available. PMID 22898002
- [Background] Dickfeld T, Kato R, Zviman M, Lai S, Meininger G, Lardo AC, Roguin A, Blumke D, Berger R, Calkins H, Halperin H. Characterization of radiofrequency ablation lesions with gadolinium-enhanced cardiovascular magnetic resonance imaging. J Am Coll Cardiol. 2006 Jan 17;47(2):370-8. doi: 10.1016/j.jacc.2005.07.070. PMID 16412863
- [Background] Lardo AC, McVeigh ER, Jumrussirikul P, Berger RD, Calkins H, Lima J, Halperin HR. Visualization and temporal/spatial characterization of cardiac radiofrequency ablation lesions using magnetic resonance imaging. Circulation. 2000 Aug 8;102(6):698-705. doi: 10.1161/01.cir.102.6.698. PMID 10931812
- [Background] Ranjan R, Kholmovski EG, Blauer J, Vijayakumar S, Volland NA, Salama ME, Parker DL, MacLeod R, Marrouche NF. Identification and acute targeting of gaps in atrial ablation lesion sets using a real-time magnetic resonance imaging system. Circ Arrhythm Electrophysiol. 2012 Dec;5(6):1130-5. doi: 10.1161/CIRCEP.112.973164. Epub 2012 Oct 15. PMID 23071143
- [Background] Ranjan R, Kato R, Zviman MM, Dickfeld TM, Roguin A, Berger RD, Tomaselli GF, Halperin HR. Gaps in the ablation line as a potential cause of recovery from electrical isolation and their visualization using MRI. Circ Arrhythm Electrophysiol. 2011 Jun;4(3):279-86. doi: 10.1161/CIRCEP.110.960567. Epub 2011 Apr 14. PMID 21493875
- [Background] Ganesan AN, Selvanayagam JB, Mahajan R, Grover S, Nayyar S, Brooks AG, Finnie J, Sunnarborg D, Lloyd T, Chakrabarty A, Abed HS, Sanders P. Mapping and ablation of the pulmonary veins and cavo-tricuspid isthmus with a magnetic resonance imaging-compatible externally irrigated ablation catheter and integrated electrophysiology system. Circ Arrhythm Electrophysiol. 2012 Dec;5(6):1136-42. doi: 10.1161/CIRCEP.112.974436. Epub 2012 Oct 16. PMID 23074322
- [Background] Vergara GR, Vijayakumar S, Kholmovski EG, Blauer JJ, Guttman MA, Gloschat C, Payne G, Vij K, Akoum NW, Daccarett M, McGann CJ, Macleod RS, Marrouche NF. Real-time magnetic resonance imaging-guided radiofrequency atrial ablation and visualization of lesion formation at 3 Tesla. Heart Rhythm. 2011 Feb;8(2):295-303. doi: 10.1016/j.hrthm.2010.10.032. Epub 2010 Oct 27. PMID 21034854
- [Background] Nordbeck P, Beer M, Kostler H, Ladd ME, Quick HH, Bauer WR, Ritter O. Cardiac catheter ablation under real-time magnetic resonance guidance. Eur Heart J. 2012 Aug;33(15):1977. doi: 10.1093/eurheartj/ehs139. Epub 2012 Jun 7. No abstract available. PMID 22677138
- [Background] Ozgun M, Maintz D, Bunck AC, Monnig G, Eckardt L, Wasmer K, Heindel W, Botnar RM, Kirchhof P. Right atrial scar detection after catheter ablation: Comparison of 2D and high spatial resolution 3D-late enhancement magnetic resonance imaging. Acad Radiol. 2011 Apr;18(4):488-94. doi: 10.1016/j.acra.2010.12.004. Epub 2011 Jan 28. PMID 21277233
- [Background] Arujuna A, Karim R, Caulfield D, Knowles B, Rhode K, Schaeffter T, Kato B, Rinaldi CA, Cooklin M, Razavi R, O'Neill MD, Gill J. Acute pulmonary vein isolation is achieved by a combination of reversible and irreversible atrial injury after catheter ablation: evidence from magnetic resonance imaging. Circ Arrhythm Electrophysiol. 2012 Aug 1;5(4):691-700. doi: 10.1161/CIRCEP.111.966523. Epub 2012 May 31. PMID 22652692
- [Background] Kiringoda R, Thurm AE, Hirschtritt ME, Koziol D, Wesley R, Swedo SE, O'Grady NP, Quezado ZM. Risks of propofol sedation/anesthesia for imaging studies in pediatric research: eight years of experience in a clinical research center. Arch Pediatr Adolesc Med. 2010 Jun;164(6):554-60. doi: 10.1001/archpediatrics.2010.75. PMID 20530306
- [Background] Niendorf HP, Alhassan A, Geens VR, Clauss W. Safety review of gadopentetate dimeglumine. Extended clinical experience after more than five million applications. Invest Radiol. 1994 Jun;29 Suppl 2:S179-82. doi: 10.1097/00004424-199406001-00059. No abstract available. PMID 7928222
- [Background] Haustein J, Laniado M, Niendorf HP, Louton T, Beck W, Planitzer J, Schoffel M, Reiser M, Kaiser W, Schorner W, et al. Triple-dose versus standard-dose gadopentetate dimeglumine: a randomized study in 199 patients. Radiology. 1993 Mar;186(3):855-60. doi: 10.1148/radiology.186.3.8430199.
- [Background] Niendorf HP, Dinger JC, Haustein J, Cornelius I, Alhassan A, Clauss W. Tolerance data of Gd-DTPA: a review. Eur J Radiol. 1991 Jul-Aug;13(1):15-20. doi: 10.1016/0720-048x(91)90049-2. PMID 1889423
- [Background] Niendorf HP, Haustein J, Cornelius I, Alhassan A, Clauss W. Safety of gadolinium-DTPA: extended clinical experience. Magn Reson Med. 1991 Dec;22(2):222-8; discussion 229-32. doi: 10.1002/mrm.1910220212. PMID 1812350
- [Background] Niendorf HP, Haustein J, Louton T, Beck W, Laniado M. Safety and tolerance after intravenous administration of 0.3 mmol/kg Gd-DTPA. Results of a randomized, controlled clinical trial. Invest Radiol. 1991 Nov;26 Suppl 1:S221-3; discussion S232-5. doi: 10.1097/00004424-199111001-00075. No abstract available. PMID 1808134
- [Background] Dillman JR, Ellis JH, Cohan RH, Strouse PJ, Jan SC. Frequency and severity of acute allergic-like reactions to gadolinium-containing i.v. contrast media in children and adults. AJR Am J Roentgenol. 2007 Dec;189(6):1533-8. doi: 10.2214/AJR.07.2554. PMID 18029897
- [Background] Sundgren PC, Leander P. Is administration of gadolinium-based contrast media to pregnant women and small children justified? J Magn Reson Imaging. 2011 Oct;34(4):750-7. doi: 10.1002/jmri.22413. PMID 21928308
- [Background] Deo A, Fogel M, Cowper SE. Nephrogenic systemic fibrosis: a population study examining the relationship of disease development to gadolinium exposure. Clin J Am Soc Nephrol. 2007 Mar;2(2):264-7. doi: 10.2215/CJN.03921106. Epub 2007 Feb 7. PMID 17699423